CLINICAL TRIAL: NCT03806894
Title: Prospective Study Evaluating Clopidogrel Resistance in Ischemic Stroke Patients From Different Ethnicities
Brief Title: Clopidogrel Resistance in Stroke Patients From Different Ethnicities
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ziv Hospital (Other Government)
Responsible Party: Principal Investigator, Dr. Najib Dally, Director of Hematology Department, Ziv Hospital
Other Study IDs: 0112-17-ZIV
Record Dates: First submitted 2019-01-15; First posted 2019-01-16 (Actual); Last update posted 2019-07-10 (Actual); Status verified 2019-07

CONDITIONS: Clopidogrel, Poor Metabolism of; Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Jewish communities: Ashkenazi, Sephardi, Ethiopian
  Interventions: Diagnostic Test: Quantification of platelet aggregation
- Arab populations: Muslim, Christian, Druze
  Interventions: Diagnostic Test: Quantification of platelet aggregation

INTERVENTIONS:
Diagnostic Test: Quantification of platelet aggregation — Platelet aggregation will be determined by vasodilator-stimulated phosphoprotein (VASP) assay

SUMMARY:
Clopidogrel is an anti-platelet agent used to inhibit blood clots. Variation in response to clopidogrel has been reported among different population and may lead to reoccurring ischemic events. The aim of the present study is to evaluate the incidence of clopidogrel resistance in ischemic stroke patients from different ethnicities in Northern Israel and to find different strategies to overcome high platelet reactivity including clopidogrel dose adjustment or the choice of alternative agents. Quantification of platelet aggregation will be determined by vasodilator stimulated phosphoprotein (VASP) assay.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to provide written informed consent and to be compliant with protocol assessments.
2. Ages 18 and above inclusive
3. Both genders eligible for the study
4. Diagnosis of ischemic cerebrovascular event

Exclusion Criteria:

1. Pregnant patients will be excluded
2. Ages below 18
3. Patients not able to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This prospective study will be conducted in two sites (Ziv Medical Center, Safed, department of neurology, and Galilee Medical Center, Nahariya, department of neurology) on 300 patients from different ethnic backgrounds with an ischemic cerebrovascular event (ischemic stroke and TIA), treated with clopidrogel for secondary stroke prevention. The groups will consist of Jewish communities (Ashkenazi, Sephardi and Ethiopian) and Arab populations (Muslim, Christian and Druze).
  To be considered eligible to participate in this study, patients have to be able to provide signed and dated written informed consent or written assent from their relatives. Both genders aged 18 and above are eligible for this trial. Pregnant patients will be excluded.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2019-10 (Estimated); Primary Completion 2020-10 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Rates of clopidogrel resistance assessed among the different ethnicities | 6 months
Identifying of high-risk subgroups of adverse clinical outcomes | 6 to 12 months